CLINICAL TRIAL: NCT03404921
Title: Efficacy and Safety of Endoscopic Submucosal Tunnel Dissection for Superficial Esophageal Squamous Cell Carcinoma: a Prospective Multicenter Study
Brief Title: Efficacy and Safety of Endoscopic Submucosal Tunnel Dissection for Superficial Esophageal Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Tongji Hospital (Other); First Affiliated Hospital of Suzhou Medical College (Other); Shanghai Zhongshan Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, Associate Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20172066-1
Record Dates: First submitted 2018-01-13; First posted 2018-01-19 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Esophageal Superficial Mucosal Lesion
Keywords: Endoscopic submucosal dissection; Endoscopic submucosal tunnelling dissection; procedure time

STUDY DESIGN:
Masking Description: The operator only understands the operation method required by the patient and is unaware of the observation indicators
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESTD group (Experimental): Use tunnelling method during ESD operation
  Interventions: Procedure: ESTD
- ESD group (Other): Use traditional method during ESD operation
  Interventions: Procedure: ESD

INTERVENTIONS:
Procedure: ESTD — During the ESTD procedure,after marking and submucosal injection, incisions were made at both the anal and oral sides of the lesion, and the submucosa under the lesion was then dissected to create a tunnel between the distal and proximal incisions. When the endscope reached the lower incision, the distal end of the esophageal lumen could be visualized , then two lateral mucosal incisions were made, thus completing the ESD procedure.
  Arms: ESTD group
Procedure: ESD — The ESD procedure involved marking,injection,circumferential cutting, submucosal dissection.
  Arms: ESD group

SUMMARY:
To evaluate the efficacy and safety profile of endoscopic submucosal tunnel dissection for superficial esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This multicenter, prospective, randomized, controlled study aims to evaluate the efficacy and safety of the tunnel technique in ESD of superficial esophageal squamous cell carcinoma (ESCC). Specifically the tunnel technique would be compared to conventional method on the procedure time and the muscular layer injury rate in patients scheduled for ESD with indication of ESCC.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years;
* Biopsy confirmed early esophageal cancer and high-grade intraepithelial neoplasia (HGIN)which were eligible for conventional ESD indications;
* Suspected localized mucosal lesions detected by endoscopy.

Exclusion Criteria:

* Malignancy or other advanced disease with a life expectancy of < 6 months as judged by the investigator.
* The ASA classification of physical status ≥ 4 as judged by the investigator.
* Severe hepatic disease or renal disease
* Ability to understand and the willingness to sign a written informed consent document.
* Major cardiovascular event at enrollment or within 3 months prior to enrollment such as stroke, myocardial infarction, or hospitalization for treatment of unstable angina pectoris as judged by the investigator.
* Haemorrhagic disorder.
* Patients who had a history of esophagectomy or a recurrent lesion.
* Planned treatment with: warfarin (including other vitamin K antagonists), cisapride,phenytoin, atazanavir, nelfinavir, digoxin, methotrexate, clopidogrel, tacrolimus,theophylline, lidocaine, nifedipine.
* Pregnancy, planned pregnancy or lactation. Women of childbearing potential must use reliable and medically accepted methods of birth control, as judged by the investigator.
* Known or suspected alcohol, drug or medication abuse.
* Any condition associated with poor compliance as judged by the investigator.
* Participation in any study involving administration of an investigational product or device within the preceding 14 days prior to enrollment.
* Involvement in the planning and conduct of the study. Previous enrollment in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The procedure time | day 1
  Procedure time was defined as the time from marking of the lesion until complete removal of the specimen,including hemostasis.

SECONDARY OUTCOMES:
The rate of bleeding during operation | day 1
  The hemorrhage observed during the operation
The rate of injury to the muscular layer | day 1
  The injury to the muscular layer observed during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, Principal Investigator — Xijing Hospital of Digestive Disease
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Fan X, Wu Q, Li R, Chen W, Xie H, Zhao X, Zhu S, Fan C, Li J, Liu M, Liu Z, Han Y. Clinical benefit of tunnel endoscopic submucosal dissection for esophageal squamous cancer: a multicenter, randomized controlled trial. Gastrointest Endosc. 2022 Sep;96(3):436-444. doi: 10.1016/j.gie.2022.04.016. Epub 2022 Apr 22. PMID 35461890